CLINICAL TRIAL: NCT02973464
Title: The Strategy in the Prevention of Renal Post-transplant Cytomegalovirus Infection Among Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Ding Xiaoming, Director of renel transplant departmet, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2016LSK-25
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Renal Transplant Recipients
MeSH Terms: interventions — Valganciclovir; Ganciclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Valganciclovir 900mg a day: Valganciclovir 900mg tablet by mouth begin within 10 days after renal transplant，once a day till to Day 100 posttransplant.
  Interventions: Drug: Valganciclovir
- Valganciclovir 450mg a day: Valgancigclovir 450 mg tablet by mouth begin within 10 days after renal transplant，once a day till to Day 100 posttransplant.
  Interventions: Drug: Valganciclovir
- Ganciclovir: Ganciclovir 5mg/kg fluids by intravenous after renal transplant，once a day for the first 14 days；and than sequential Ganciclovir 1g tablet by mouth，third a day till to Day 100 posttransplant.
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Oral at a dose of 450mg or 900mg per day begin within 10 days till to Day 100 posttransplant
  Other Names: Valcyte; Valin ganciclovir; VGC
  Groups: Valganciclovir 450mg a day; Valganciclovir 900mg a day
Drug: Ganciclovir — intravenous GCV 5mg/kg/d after renal transplantation for the first 14 days, and then oral GCV 1g 3 times daily till to Day 100 posttransplant.
  Other Names: Cymevene; GCV
  Groups: Ganciclovir

SUMMARY:
This study evaluates the safety and availability of oral valganciclovir(VGC) at the does of 450mg daily begin within 10 days after renal transplantation, and till to Day 100 posttransplant. Compare to the guidelines for effective antiviral prophylaxis, the investigators divide these patients into three groups in random. One third will oral VGC 450mg daily as mentioned above; one third will oral VGC 900mg daily; and the other one third will intravenous GCV 5mg/kg daily within the first 14 days posttransplant, and continue to oral GCV 1g 3 times daily till to Day 100 posttransplant; with does adjusted per renal function for all agents.

DETAILED DESCRIPTION:
Human Cytomegalovirus(CMV), a kind of β-hepersvirus, which is a common opportunistic pathogen. The ubiquity of CMV infection in human beings had been verified; and the CMV-IgG seropositive rate is 97% among healthy population, most of them are at the state of latent infection. When immunosuppressed, such as for renal transplant recipients, the incidence of CMV infection and disease increase obviously. The posttransplant CMV infection would induce allgraft rejection, impact on allgraft and recipients survival, as well as contribute to the serious complications.Many studies show that giving effective antivirus drugs after transplantation is benifit to recipients.

Nowadays,the strategy of intravenous GCV GCV 5mg/kg daily or oral GCV 1g 3 times daily, which is the recommended treatment for CMV disease posttransplantation.Resent date show that VGC is an oral prodrug of GCV. When VGC is absorbed in the intestinal wall and liver, it is rapidly metabolized to ganciclovir. As a contemporary study, IV GCV 5mg/kg/day will approach to a similar area under the curve to VGC 900mg daily. The bioavailability of ganciglovir from valganciclovir is 10 times of GCV by oral. For recipients, oral therapy is more safety and convinient, so that it will reduce frequent hospitalizations. As many researches, it is indicated that oral VGC 450mg daily can also reduce the adverse events resulting from posttransplant CMV infection, there is no significantly statistic differences when compared with oral VGC 900mg daily. Simultaneously, lower dose could decrease the risk of leukopenia and ease the burden for recipients.

This study is a single-center, prospective, observational, corhort study. According to the inclusion and exclusion criteria, the investigators will recruit 450 patients. And every one will be followed up for at least 12 months unless death or graft loss, the specific duration is at baseline, weekly within the first 3 months posttransplantation, month 4, month 5, month 6, month 9, and month 12. Recipients will be followed for CMV-DNA, CMV-pp65, CMV antigenemia, blood routine test, urinalysis, liver function, renal fuction and the chest X-ray films. Inverstigators should collect the date of recipient as below: general conditions, such as age, sex, weight and so on; primary reason for transplant; donor/recipient CMV serostatus; biopsy-prove acute rejection; opportunistic infections; NODAT; etc. And Chi-square or Fisher's exact test will be used as appropriate to compare categorical variables, and it is considered as statistically significant when the 2-sided P-value<0.05. Definitively, conclusion will be come out to verify the safety and availability of our protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1.65 years old>=Age>=18 years old, male or female
* 2.Renal transplantation first time
* 3.CMV serology donor-positive(D+) or recipient-positive(R+) renal transplant recipients

Exclusion Criteria:

* 1.Those who are allergic or resistant to Acyclovir, Valaciclovir, Ganciclovir, Valganciclovir
* 2.HIV, hepatitis B or hepatitis C patients
* 3.Not in pregnancy or lactation, pregnancy test was negative, and promise not to be pregnancy during treatment
* 4.Male with a pregnant partner; or lactation
* 5.Suspected CMV disease at enrolment
* 6.Use of anti-CMV therapy within 30 days prior to study
* 7.Multiple organ transplantation
* 8.Uncontrolled diarrhea or evidence of malabsorption
* 9.Liver function tests>3 times the upper level of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
incidence of CMV infection and disease | within the first 1 year after renal transplant

SECONDARY OUTCOMES:
incidence of CMV infection and disease | within the first 3 and 6 months after renal transplant respectively
GCV-resistant CMV infection | within the first 1 year after renal transplant
mean estimated renal function, allograft survival and patient survival | within the first 1 year after renal transplant
incidence of acute rejection | within the first 1 year after renal transplant
other opportunistic infections | within the first 1 year after renal transplant
adverse events, such as NODAT | within the first 1 year after renal transplant

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming D Ding, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomasec P, Braud VM, Rickards C, Powell MB, McSharry BP, Gadola S, Cerundolo V, Borysiewicz LK, McMichael AJ, Wilkinson GW. Surface expression of HLA-E, an inhibitor of natural killer cells, enhanced by human cytomegalovirus gpUL40. Science. 2000 Feb 11;287(5455):1031. doi: 10.1126/science.287.5455.1031. PMID 10669413
- [Background] Retiere C, Prod'homme V, Imbert-Marcille BM, Bonneville M, Vie H, Hallet MM. Generation of cytomegalovirus-specific human T-lymphocyte clones by using autologous B-lymphoblastoid cells with stable expression of pp65 or IE1 proteins: a tool to study the fine specificity of the antiviral response. J Virol. 2000 May;74(9):3948-52. doi: 10.1128/jvi.74.9.3948-3952.2000. PMID 10756006
- [Background] Zheng Q, Tao R, Gao H, Xu J, Shang S, Zhao N. HCMV-encoded UL128 enhances TNF-alpha and IL-6 expression and promotes PBMC proliferation through the MAPK/ERK pathway in vitro. Viral Immunol. 2012 Apr;25(2):98-105. doi: 10.1089/vim.2011.0064. PMID 22486303
- [Background] Rubin RH. Infectious disease complications of renal transplantation. Kidney Int. 1993 Jul;44(1):221-36. doi: 10.1038/ki.1993.234. No abstract available. PMID 8394951
- [Background] Schmaldienst S, Horl WH. Bacterial infections after renal transplantation. Nephron. 1997;75(2):140-53. doi: 10.1159/000189523. No abstract available. PMID 9041533
- [Background] Streblow DN, Orloff SL, Nelson JA. Acceleration of allograft failure by cytomegalovirus. Curr Opin Immunol. 2007 Oct;19(5):577-82. doi: 10.1016/j.coi.2007.07.012. Epub 2007 Aug 22. PMID 17716883
- [Background] Szczepura A, Westmoreland D, Vinogradova Y, Fox J, Clark M. Evaluation of molecular techniques in prediction and diagnosis of cytomegalovirus disease in immunocompromised patients. Health Technol Assess. 2006 Apr;10(10):1-176. doi: 10.3310/hta10100. PMID 16595079
- [Background] Bendiksen S, Van Ghelue M, Rekvig OP, Gutteberg T, Haga HJ, Moens U. A longitudinal study of human cytomegalovirus serology and viruria fails to detect active viral infection in 20 systemic lupus erythematosus patients. Lupus. 2000;9(2):120-6. doi: 10.1191/096120300678828118. PMID 10787009
- [Background] Zhou L, Fan J, Zheng SS, Ma WH. Prevalence of human cytomegalovirus UL97 D605E mutation in transplant recipients in China. Transplant Proc. 2006 Nov;38(9):2926-8. doi: 10.1016/j.transproceed.2006.08.161. PMID 17112867
- [Background] Dong B, Wang Y, Wang G, Wang W, Zhou H, Fu Y. A retrospective study of cytomegalovirus pneumonia in renal transplant patients. Exp Ther Med. 2014 May;7(5):1111-1115. doi: 10.3892/etm.2014.1577. Epub 2014 Feb 24. PMID 24940395
- [Background] Meije Y, Fortun J, Len O, Aguado JM, Moreno A, Cisneros JM, Gurgui M, Carratala J, Munoz P, Montejo M, Blanes M, Bou G, Perez JL, Torre-Cisneros J, Ramos A, Pahissa A, Gavalda J; Spanish Network for Research on Infection in Transplantation (RESITRA) and the Spanish Network for Research on Infectious Diseases (REIPI). Prevention strategies for cytomegalovirus disease and long-term outcomes in the high-risk transplant patient (D+/R-): experience from the RESITRA-REIPI cohort. Transpl Infect Dis. 2014 Jun;16(3):387-96. doi: 10.1111/tid.12226. Epub 2014 May 8. PMID 24807640
- [Background] Fernandez-Ruiz M, Arias M, Campistol JM, Navarro D, Gomez-Huertas E, Gomez-Marquez G, Diaz JM, Hernandez D, Bernal-Blanco G, Cofan F, Jimeno L, Franco-Esteve A, Gonzalez E, Moreso FJ, Gomez-Alamillo C, Mendiluce A, Luna-Huerta E, Aguado JM; OPERA Study Group. Cytomegalovirus prevention strategies in seropositive kidney transplant recipients: an insight into current clinical practice. Transpl Int. 2015 Sep;28(9):1042-54. doi: 10.1111/tri.12586. Epub 2015 Apr 23. PMID 25864986
- [Background] Khoury JA, Storch GA, Bohl DL, Schuessler RM, Torrence SM, Lockwood M, Gaudreault-Keener M, Koch MJ, Miller BW, Hardinger KL, Schnitzler MA, Brennan DC. Prophylactic versus preemptive oral valganciclovir for the management of cytomegalovirus infection in adult renal transplant recipients. Am J Transplant. 2006 Sep;6(9):2134-43. doi: 10.1111/j.1600-6143.2006.01413.x. Epub 2006 Jun 19. PMID 16780548
- [Result] Asberg A, Humar A, Rollag H, Jardine AG, Mouas H, Pescovitz MD, Sgarabotto D, Tuncer M, Noronha IL, Hartmann A; VICTOR Study Group. Oral valganciclovir is noninferior to intravenous ganciclovir for the treatment of cytomegalovirus disease in solid organ transplant recipients. Am J Transplant. 2007 Sep;7(9):2106-13. doi: 10.1111/j.1600-6143.2007.01910.x. Epub 2007 Jul 19. PMID 17640310
- [Result] Humar A, Lebranchu Y, Vincenti F, Blumberg EA, Punch JD, Limaye AP, Abramowicz D, Jardine AG, Voulgari AT, Ives J, Hauser IA, Peeters P. The efficacy and safety of 200 days valganciclovir cytomegalovirus prophylaxis in high-risk kidney transplant recipients. Am J Transplant. 2010 May;10(5):1228-37. doi: 10.1111/j.1600-6143.2010.03074.x. Epub 2010 Mar 26. PMID 20353469
- [Result] Tu PT, Shu KH, Cheng CH, Chen CH, Yu TM, Chuang YW, Huang ST, Tsai SF, Cheng CY, Wu MJ. Universal valganciclovir prophylaxis significantly reduces episodes of first-year cytomegalovirus disease and biopsy-proven acute rejection in kidney transplant recipients. Transplant Proc. 2014;46(2):574-7. doi: 10.1016/j.transproceed.2013.11.115. PMID 24656016
- [Result] Stevens DR, Sawinski D, Blumberg E, Galanakis N, Bloom RD, Trofe-Clark J. Increased risk of breakthrough infection among cytomegalovirus donor-positive/recipient-negative kidney transplant recipients receiving lower-dose valganciclovir prophylaxis. Transpl Infect Dis. 2015 Apr;17(2):163-73. doi: 10.1111/tid.12349. Epub 2015 Feb 6. PMID 25661673